CLINICAL TRIAL: NCT01653067
Title: A Phase II Trial to Evaluate the Safety, Feasibility and Efficacy of a Salvage Therapy Consisting of Temsirolimus Added to the Standard Therapy R-DHAP for the Treatment of Patients With Relapsed or Refractory DLBCL - the STORM Trial
Brief Title: STORM: Temsirolimus, Rituximab and DHAP for Relapsed and Refractory Diffuse Large B-cell Lymphoma
Acronym: STORM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mathias Witzens-Harig (Other)
Collaborators: Johannes Gutenberg University Mainz (Other); Technical University of Munich (Other); Ludwig-Maximilians - University of Munich (Other); University Hospital Ulm (Other); University Hospital Erlangen (Other); Charite University, Berlin, Germany (Other); University Hospital Freiburg (Other); Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Sponsor-Investigator, Mathias Witzens-Harig, PD Dr. med. Mathias Witzens-Harig, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STORM-2011; 2011-001491-20 (EudraCT Number)
Record Dates: First submitted 2012-07-17; First posted 2012-07-30 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Non Hodgkin´s Lymphoma; Diffuse Large B-Cell Lymphoma; Aggressive Lymphoma; Aggressive Non Hodgkin´s Lymphoma; NHL; aNHL; Temsirolimus; Torisel; Relapsed Non Hodgkin´s Lymphoma; Relapsed Diffuse Large B-Cell Lymphoma; aggressive NHL; B-NHL; aggressive B-NHL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Rituximab; temsirolimus; dexamethasone acetate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab, Temsirolimus, DHAP, intravenous (Experimental): This is a multicenter, open label, single arm, phase II study. There will be no placebo usage within this trial. In the part I, dose escalation part, of this trial 6 patients will be included in each dose level. There will be 4 cohorts, administering up to a maximum of 4 cycles 25 mg, 50 mg, 75mg or 100mg Temsirolimus in combination with Rituximab and DHAP.
  Treatment regimen part I:
  Part I - Cohort A, B, C, D, X Temsirolimus 25 (A), 50 (B), 75 (C),100 (D) or 15 (X) mg, Day 1, 8, Rituximab (375 mg/m² day 2) Dexamethasone 40mg day 3-6 Cisplatine 100 mg/m² day 3 Cytarabine 2x2 g/m² day 4
  ...repeat day 22, up to a maximum of 4 cycles
  In the part II of the trial 40 patients will be included to receive the full target dose, established within the part I of the study.
  Interventions: Drug: Rituximab, Temsirolimus, DHAP, intravenous

INTERVENTIONS:
Drug: Rituximab, Temsirolimus, DHAP, intravenous — Maximum tolerated dose of Temsirolimus Rituximab (375 mg/m²) Dexamethasone (120 mg) Cisplatin (100mg/m²) Cytarabine (2x2g/m²))
  Other Names: Temsirolimus-R-DHAP; Torisel; MabThera; Fortecortin; ARA-C; ARA-cell; Depocyte; R-DHAP; Rituximab-DHAP; Temsirolimus,Rituximab,Dexamethasone,Cisplatine,Cytarabine; Temsirolimus-Rituximab-DHAP

SUMMARY:
The STORM-trial consists of two parts. In the part I (dose escalation of Temsirolimus) the primary objective is to establish a maximum tolerated dose of Temsirolimus in combination with Rituximab and DHAP. Secondary objective is to prove ability to mobilize stem cells in patients scheduled to high dose therapy.

In the part II (full target dose) the primary objective is to evaluate the ORR in patients with relapsed diffuse large B cell lymphoma (DLBCL). The secondary objective is to evaluate progression free survival (PFS), overall survival (OS) and Toxicity.

DETAILED DESCRIPTION:
This is a multicenter, open label, single arm, phase II study. There will be no placebo usage within this trial. In the part I, dose escalation part, of this trial 6 patients will be included in each dose level. There will be 4 cohorts, administering up to a maximum of 4 cycles 25 mg, 50 mg, 75mg or 100mg Temsirolimus in combination with Rituximab and DHAP.

Treatment regimen part I:

Part I - Cohort A, B, C, D, X Temsirolimus 25 (A), 50 (B), 75 (C),100 (D) or 15 (X) mg, Day 1, 8, Rituximab (375 mg/m² day 2) Dexamethasone 40mg day 3-6 Cisplatine 100 mg/m² day 3 Cytarabine 2x2 g/m² day 4

...repeat day 22, up to a maximum of 4 cycles In part I, after inclusion of 6 patients, each patient has to receive at least 1 complete cycle w/o dose limiting toxicity until the enrollment into the next cohort can be initiated.

In the part II of the trial 40 patients will be included to receive the full target dose, established within the part I of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven diagnosis of diffuse large cell B-cell lymphoma (DLBCL) according to the World Health Organization classification.
* Documented relapse or progression following at least one treatment but a maximum of 2 prior treatments. Prior treatment must have included at least 3 cycles of anthracycline containing chemotherapy (e.g. CHOP-like)
* Any of the following: at least 1 measurable tumor mass (>1.5 cm x >1.0 cm), involvement of any organ or bone marrow infiltration
* Subjects 18 years or older
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Adequate bone marrow reserve: Platelets of at least 75000/µl, absolute neutrophil count at least 1500/µl
* Alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN); Aspartate aminotransferase (AST) < 2.5 x ULN, Total bilirubin < 1.5 x ULN
* Calculated creatinine clearance (MDRD) > 70 mL/min
* Eastern Cooperative Oncology Group [ECOG] performance Status < 3
* Female subject must be postmenopausal (for at least 6 months), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study; and have a negative serum ß-hCG pregnancy test at screening

Exclusion Criteria:

* Active central nervous System lymphoma. Brain MRI is required only if clinically indicated
* Pregnancy or breast feeding women
* Lymphoma other than DLBCL
* Severe concomitant disease (e.g. uncontrolled arterial hypertension, heart failure (NYHA III-IV), uncontrolled diabetes mellitus, pulmonary fibrosis, uncontrolled hyperlipoproteinemia)
* Active uncontrolled infections including HIV-positivity, active Hep B or C
* Mental status precluding patient's compliance
* Prior treatment with Temsirolimus
* Known CD20 negativity
* Patients refractory to DHAP in a prior treatment line
* Prior autologous or allogeneic stem cell or bone marrow transplantation
* Peripheral neuropathy or neuropathic pain of Grade 2 or worse
* Diagnosed or treated for a malignancy other than NHL except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, DCIS of the breast, or other solid tumors curatively treated with no evidence of disease for >5 years
* Concurrent treatment with another investigational agent during the conduct of the trial.
* Concurrent participation in non-treatment studies is not excluded
* Known intolerance to Sirolimus or derivates, Cytarabine, Cisplatine or Rituximab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Safety, Tolerability and Efficacy of a combination therapy of Temsirolimus added to the standard therapy, Rituximab and DHAP (Cytarabine, Cisplatine, Dexamethasone) | 09-2012 to 06-2018 (up to six years)
  In the part I (dose escalation of Temsirolimus) the primary objective is to establish a maximum tolerated dose of Temsirolimus in combination with Rituximab and DHAP.

SECONDARY OUTCOMES:
Safety, Tolerability and Efficacy of a combination therapy of Temsirolimus added to the standard therapy, Rituximab and DHAP (Cytarabine, Cisplatine, Dexamethasone) | 09-2012 to 06-2018 (up to six years)
  In the part I (dose escalation of Temsirolimus) secondary objective is to prove ability to mobilize stem cells in patients scheduled to high dose therapy.
Safety, Tolerability and Efficacy of a combination therapy of Temsirolimus added to the standard therapy, Rituximab and DHAP (Cytarabine, Cisplatine, Dexamethasone) | 09-2012 to 06-2018 (up to six years)
  In the part II (full target dose) the secondary objective is to evaluate Progression Free Survival
Safety, Tolerability and Efficacy of a combination therapy of Temsirolimus added to the standard therapy, Rituximab and DHAP (Cytarabine, Cisplatine, Dexamethasone) | 09-2012 to 06-2018 (up to six years)
  In the part II (full target dose) the secondary objective is to evaluate Overall Survival
Safety, Tolerability and Efficacy of a combination therapy of Temsirolimus added to the standard therapy, Rituximab and DHAP (Cytarabine, Cisplatine, Dexamethasone) | 09-2012 to 06-2018 (up to six years)
  In the part II (full target dose) the secondary objective is to evaluate Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Witzens-Harig, MD, Principal Investigator — University Hospital of Heidelberg, Department 5 Hematology, Oncology, Rheumatology, Im Neuenheimer Feld 410, 69120 Heidelberg, Germany
Locations (9):
- Germany (9):
  - University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - University of Heidelberg Hospital, Heidelberg, Baden-Wurttemberg
  - University Hospital Ulm, Ulm, Baden-Wurttemberg
  - University Hospital Erlangen, Erlangen, Bavaria
  - Ludwig-Maximilians-University of Munich, Munich, Bavaria
  - Technische Universität München, Munich, Bavaria
  - Johann Wolfgang Goethe University Hospitals, Frankfurt, Frankfurt am Main, Hesse
  - Johannes Guttenberg University Mainz, Mainz, Rhineland-Palatinate
  - Charité University Berlin, Berlin, State of Berlin

REFERENCES:
- [Derived] Witzens-Harig M, Memmer ML, Dreyling M, Hess G. A phase I/II trial to evaluate the safety, feasibility and activity of salvage therapy consisting of the mTOR inhibitor Temsirolimus added to standard therapy of Rituximab and DHAP for the treatment of patients with relapsed or refractory diffuse large cell B-Cell lymphoma - the STORM trial. BMC Cancer. 2013 Jun 25;13:308. doi: 10.1186/1471-2407-13-308. PMID 23799873